CLINICAL TRIAL: NCT06416605
Title: Tooth Shell Versus Bone Shell Technique For Horizontal Maxillary Alveolar Ridge Augmentation
Brief Title: Autogenous Tooth Graft for Ridge Augmentation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elsheikh, Assistant Professor of Oral and Maxillofacial Surgery, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A03030123
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dental Implant
MeSH Terms: interventions — Alveolar Ridge Augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Horizontal bone augmentation will be done by bone shell technique
  Interventions: Procedure: Maxillary Alveolar Ridge Augmentation
- group B (Experimental): Horizontal bone augmentation will be done by autogenous tooth shell technique
  Interventions: Procedure: Maxillary Alveolar Ridge Augmentation

INTERVENTIONS:
Procedure: Maxillary Alveolar Ridge Augmentation — using tooth graft or bone graft to increase alveolar ridge width to be able to insert dental implant

SUMMARY:
This study is designed to evaluate the clinical and radiographical outcome of tooth shell for alveolar ridge reconstruction in maxilla as an alternative to traditional autologous bone shell graft.

DETAILED DESCRIPTION:
twenty eight patients with one or two maxillary extracted teeth in need for horizontal bone augmentation and implant placement will be selected from the outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University patients will be divided into two equal groups:

• Group I: Horizontal bone augmentation will be done by bone shell technique.

• Group II: Horizontal bone augmentation will be done by autogenous tooth shell technique.

Evaluation:

A-Clinical evaluation:

* All patients were followed up on a weekly basis for the first postoperative month, then monthly for the rest of the postoperative period (6months) until implantation.
* The patients were evaluated regarding pain, edema and hematoma at recipient and donor sites as well as healing of the mucosa.
* A neurosensory evaluation was carried out at each clinical check up by asking the patient if there were any areas of hypoesthesia, numbness or tingling in the lower lip and chin at the side of the donor site.

B-Radiographic evaluation

•Cone beam computed tomography (CBCT) were made immediately and 6 months post-operative to assess the alveolar bone in all three planes of space before implant placement. According to the measurements obtained from CBCT, appropriate implant size and length will be chosen and placed 6 months postoperative after removal of the micro screws.

Radiographic analysis:

Linear measurements of alveolar bone width were taken using CBCT scan at three stages; prior to grafting (T0) and immediately (T1), and 4 months post grafting (T2). Then three horizontal alveolar width measurements (crestal, middle and apical) were recorded at T0, T2 and T1. The measurement was performed with fixed points each time, the buccolingual width was measured at different levels. At the bone crest, 3mm from the bone crest and 6mm from the bone crest. The measurements were tabulated for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

- 1- One or two maxillary extracted teeth with crestal bone width of 4 mm or less.

2- Age ranging from 18_50 years 3- 3- Adequate oral hygiene. 4- Non smoking patients. 5-Free from any pathological lesions related to the tooth to be extracted. 6- Physically fit to withstand the whole procedure.

Exclusion Criteria:

* 1- Active infection in the site to be treated. 2- Patients on chemotherapy or radiotherapy. 3- Alcohol or drug abuse. 4- Patients who have systemic disorders that interfere with bone healing {uncontrolled diabetes mellitus, autoimmune disease,

  * etc.} 5- Pregnancy. 6- Patients with bone disease. 7- Patients with parafunctional habits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
horizontal alveolar width measurements | 6 months
  Cone beam computed tomography (CBCT) were made immediately and 6 months post-operative to assess the alveolar bone in all three planes of space before implant placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt

REFERENCES:
- [Derived] Awad KAI, Tawik MA, Hussein MM, El-Farag SAA, Sameaa SESA. Tooth shell versus bone shell technique for horizontal maxillary alveolar ridge augmentation. BMC Oral Health. 2025 Apr 25;25(1):642. doi: 10.1186/s12903-025-05940-4. PMID 40281533